CLINICAL TRIAL: NCT06626477
Title: Intra-Nasal Mechanical Stimulation (INMEST) as a Potential Treatment Method for Sjogren's Syndrome (SS) - a Prospective, Double-Blind, Randomized Pilot Study To Evaluate the Safety and Performance of the Walther System
Brief Title: Intra-Nasal Mechanical Stimulation (INMEST) as a Potential Treatment Method for Sjogren's Syndrome (SS)
Acronym: A-SS-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abilion Medical Systems AB (Industry)
Collaborators: Insamlingsstiftelsen för främjande av forskning avseende INMEST (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-SS-001; CIV-24-05-047403 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Sjogren Syndrome
Keywords: INMEST; Abilion
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: During the first half (6 weeks) the subjects receive either active or sham treatment (randomized). During the final half (6 weeks) all subjects receive active treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Manufacturer, Monitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (6 weeks) + Active (6 weeks) (Experimental): Randomized, double-blinded, active treatment for 6 weeks, then 6 weeks of unblinded active treatment.
  Interventions: Device: Intra nasal mechanical stimulation treatment (INMEST)
- Sham (6 weeks) + Active (6 weeks) (Sham Comparator): Randomized, double-blinded, sham treatment for 6 weeks, then 6 weeks of unblinded active treatment.
  Interventions: Device: Intra nasal mechanical stimulation treatment (INMEST); Device: Sham (No Treatment)

INTERVENTIONS:
Device: Intra nasal mechanical stimulation treatment (INMEST) — The treatment is performed with the Walther System manufactured by Abilion Medical Systems AB.
  Other Names: INMEST
Device: Sham (No Treatment) — A modified Walther System not delivering active treatment manufactured by Abilion Medical Systems AB.
  Arms: Sham (6 weeks) + Active (6 weeks)

SUMMARY:
The purpose of the study is to investigate the effect and safety of the Walther System delivering INMEST (intranasal mechanical stimulation) on people with Sjogren's syndrome. A total of 30 subjects are planned to be enrolled and randomized to either use an active device or a sham device for the first 6 weeks. During the last 6 weeks all subjects will receive active treatment. The treatments are self-administered by the subject at home, three times a week and 10 minutes per nostril.

Subjects will:

* Use an active or sham device at home 3 times per week for six weeks.
* All subjects will then get an active device for use another six weeks.
* Visit the clinic every third week for measurements and checkups.
* Keep a diary of the treatments and potential problems.

DETAILED DESCRIPTION:
Clinical investigation purpose and background ----- In this investigation the intended purpose of the investigational device, the Walther System, is to deliver intranasal mechanical stimulation (INMEST) for symptom relief in cases of Sjogren's syndrome, and the treatment is self-administered at home.

Sjogren's syndrome is a chronic disorder of the immune system that usually affects the mucous membranes and moisture-secreting glands of the eyes and mouth. The two most common symptoms of Sjogren's Syndrome are dry eyes and a dry mouth. The prevalence has been reported to be 0.06% and the disease mostly affect women and people over 40. There are currently no treatment options for Sjogren's syndrome other than relieving symptoms resulting in medications that decrease eye inflammation, increase saliva production, and/or suppress the immune system.

Design of clinical investigation

-----

This is a randomized, double-blinded, single centre, pilot study with a total of 30 study subjects, from 18 years of both genders. Randomization of study subjects is done in permuted blocks and the subjects are randomized to either one of two groups of equal size receiving either:

A. treatment with the investigational device (active) B. treatment with comparator device (sham/control) After half the treatment time all subjects are given a new investigational device that is active, thus all subjects will receive active treatment.

After enrolment in the study, including the informed consent procedure, and the subsequent randomization process, study subjects are assigned to either an investigational device treatment (group A) or a comparator treatment group (group B). After an initial demonstration of the device (comparator or investigational device), study subjects will be given the device to be used for self-administration at home, 3 days a week, 10 minutes per nasal cavity (i.e. a total of 20 minutes per treatment session), for a total treatment period of 12 weeks (i.e., a total of 36 treatment sessions). After 6 weeks all subjects, irrespective of group, will exchange their device for an investigational device, thus all subjects will receive active treatment for the last 6 weeks.

Clinic visits with measurements are scheduled at baseline followed at visits after 3, 6, 9, and 12 weeks when end of treatment is reached. Every visit after baseline should be made within a time window of -3 days to +10 days. Subjects are instructed not to perform any treatments with the device 12 hours prior visiting the clinic.

During the study period, both patients' reported symptoms and objective measurements will be collected. An analysis will also be made of compliance with the prescribed treatment and the safety of the investigational medical device will be evaluated through analysis of reported adverse events and device deficiencies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at inclusion date
2. Schirmer's test ≤ 5 mm for both eyes
3. NIBUT ≤ 10 s for both eyes
4. Previous positive result of blood test for sample anti-Ro (SS-A) or anti-La (SS-B), as indicated by medical record or lab result shown by the subject.
5. The study subject reports having understood and have signed the Informed Consent Form (ICF) and is willing to comply with all investigation visits and assessments.
6. Women of childbearing potential must agree to use a reliable, medically approved form of contraception during the study participation until end of study.
7. Anticipated compliance with prescribed treatment and follow-up.

Exclusion Criteria:

1. Recently (12 months prior enrolment) undergone nasal, sinus, or ocular surgery.
2. Presence of an ocular or respiratory condition that could affect the study parameters such as active ocular infection/inflammation, glaucoma, diabetic retinopathy, or upper respiratory tract infection per the Investigator's judgement.
3. The study subject has a cognitive incapacity or language barrier precluding adequate understanding or cooperation.
4. Any severe diseases interfering with the performance, evaluation, and outcome of the clinical evaluation.
5. The study subject is considered by the Investigator to be unsuitable to participate in the investigation for any other reason.
6. Previous (within 30 days prior to enrolment) and concurrent treatment with another investigational drug/s or device/s.
7. Subject is pregnant or lactating or planning to get pregnant during the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-07-19 (Actual); Study Completion 2025-07-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean Schirmer's test at six weeks | From enrollment to week 6
  Change in mean tear production using Schirmer's test comparing active treatment (active) vs sham treatment (control) evaluated at baseline (Day 0) and week 6 (Day 42) comparing active and sham treatment.

SECONDARY OUTCOMES:
Adverse Events | From enrollment to the end of treatment at 12 weeks
  Number of treatment related Adverse Events/Adverse Device Effects/Serious Adverse Events/Serious Adverse Device Effects and Unanticipated Serious Adverse Device Effects when using the Walther System.
Device Deficiencies | From enrollment to the end of treatment at 12 weeks
  Number of Walther System Device Deficiencies.
Change from baseline in the mean Best-Corrected Visual Acuity (BCVA) at six weeks | From enrollment to week 6
  Change in mean Best-Corrected Visual Acuity (BCVA) using a Snellen equivalent chart evaluated at baseline (Day 0) and week 6 (Day 42) comparing active and sham treatment.
Change from baseline in the mean Non-invasive Break-Up (NIBUT) time at six weeks | From enrollment to week 6
  Change in mean Non-invasive Break-Up time (NIBUT) evaluated at baseline (Day 0) and week 6 (Day 42) comparing active and sham treatment.
Change from baseline in the mean Fluorescein Eye Stain Test at six weeks | From enrollment to week 6
  Change in Fluorescein Eye Stain Test evaluated at baseline (Day 0) and week 6 (Day 42) comparing active and sham treatment.
Change from baseline in Matrix Metalloproteinase-9 (MMP-9) at six weeks | From enrollment to week 6
  Change in Matrix Metalloproteinase-9 (MMP-9) evaluated at baseline (Day 0) and week 6 (Day 42) comparing active and sham treatment.
Change from baseline in the mean salivary flow rate time at six weeks | From enrollment to week 6
  Change in mean salivary flow rate evaluated at baseline (Day 0) and week 6 (Day 42) comparing active and sham treatment.
Change from baseline in the mean EULAR Sjogrens Syndrome Patient Reported Index (ESSPRI) at six weeks | From enrollment to week 6
  Self-experienced change in mean EULAR Sjogrens Syndrome Patient Reported Index (ESSPRI) evaluated at baseline (Day 0) and week 6 (Day 42) comparing active and sham treatment.
Change from baseline in the mean Ocular Surface Disease Index (OSDI) at 6 weeks | From enrollment to week 6
  Self-experienced change in Ocular Surface Disease Index (OSDI) evaluated at baseline (Day 0) and week 6 (Day 42) comparing active and sham treatment.
Change in the mean Schirmers test between six and twelve weeks active treatment | From enrollment to week 12 (Active) and from week 7 to 12 (Control)
  Change in mean tear production using Schirmer's test comparing active group (12 weeks) with control group (6 last weeks of active treatment).
Change in the mean Best-Corrected Visual Acuity (BCVA) between six and twelve weeks active treatment | From enrollment to week 12 (Active) and from week 7 to 12 (Control)
  Change in Best-Corrected Visual Acuity (BCVA) using a Snellen equivalent chart comparing active group (12 weeks) with control group (6 last weeks of active treatment).
Change in the mean Fluorescein Eye Stain Test between six and twelve weeks active treatment | From enrollment to week 12 (Active) and from week 7 to 12 (Control)
  Change in mean Fluorescein Eye Stain Test evaluated at baseline (Day 0) and week 6 (Day 42) comparing active group (12 weeks) with control group (6 last weeks of active treatment).
Change in Matrix Metalloproteinase-9 (MMP-9) between six and twelve weeks active treatment | From enrollment to week 12 (Active) and from week 7 to 12 (Control)
  Change in Matrix Metalloproteinase-9 (MMP-9) evaluated at baseline (Day 0) and week 6 (Day 42) comparing active group (12 weeks) with control group (6 last weeks of active treatment).
Change in the mean salivary flow rate time between six and twelve weeks active treatment | From enrollment to week 12 (Active) and from week 7 to 12 (Control)
  Change in mean salivary flow rate comparing active group (12 weeks) with control group (6 last weeks of active treatment).
Change in the mean EULAR Sjogrens Syndrome Patient Reported Index (ESSPRI) between six and twelve weeks active treatment | From enrollment to week 12 (Active) and from week 7 to 12 (Control)
  Self-experienced change in mean EULAR Sjogrens Syndrome Patient Reported Index (ESSPRI) comparing active group (12 weeks) with control group (6 last weeks of active treatment).
Change in the mean Ocular Surface Disease Index (OSDI) between six and twelve weeks active treatment | From enrollment to week 12 (Active) and from week 7 to 12 (Control)
  Self-experienced change in mean Ocular Surface Disease Index (OSDI) comparing active group (12 weeks) with control group (6 last weeks of active treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Källmark, PhD, Principal Investigator — Källmarkskliniken AB
Locations (1):
- Källmarkskliniken AB, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No